CLINICAL TRIAL: NCT06782555
Title: A Phase 1/2 Immunotherapy Study of Evofosfamide in Combination with Zalifrelimab and Balstilimab in Patients with Advanced Solid Malignancies
Brief Title: A Study of Evofosfamide in Combination with Zalifrelimab and Balstilimab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunoGenesis (Industry)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EVO-011
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Prostate Cancer; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Squamous Cell Carcinoma of Head and Neck; Pancreatic Neoplasms | interventions — TH 302; balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Castration-resistant prostate cancer (Experimental): Evofosfamide + zalifrelimab + balstilimab
  Interventions: Drug: Evofosfamide; Drug: Zalifrelimab; Drug: Balstilimab
- Pancreatic cancer (Experimental): Evofosfamide + zalifrelimab + balstilimab
  Interventions: Drug: Evofosfamide; Drug: Zalifrelimab; Drug: Balstilimab
- Human papilloma virus-negative squamous cell carcinoma of the head and neck (Experimental): Evofosfamide + zalifrelimab + balstilimab
  Interventions: Drug: Evofosfamide; Drug: Zalifrelimab; Drug: Balstilimab

INTERVENTIONS:
Drug: Evofosfamide — Evofosfamide administered on Days 1 and 8 of Cycles 1, 2, and 3.
Drug: Zalifrelimab — Zalifrelimab administered on Day 8 of Cycles 1, 3, and 5.
Drug: Balstilimab — Balstilimab administered every 2 weeks beginning on Day 8 of Cycle 1.

SUMMARY:
The purpose of this Phase 1/2 study is to test the overall safety, tolerability, and effectiveness of the combination investigational drugs evofosfamide, zalifrelimab, and balstilimab in treating advanced or metastatic castration-resistant prostate cancer, pancreatic cancer, and human papilloma virus (HPV)-negative squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
Tumor hypoxia can lead to poor effector T-cell penetration and immunosuppressive signaling via myeloid-derived suppressor cells, myofibroblasts, and regulatory T-cells. Disruption of these hypoxic regions within the tumor microenvironment by the hypoxia-directed cytotoxic agent evofosfamide may enhance the ability of immune checkpoint inhibitors to reject otherwise resistant solid tumors. The hypothesis tested in this study is that evofosfamide, by specifically targeting the hypoxic tumor microenvironment, may enhance the anti-tumor effects of the immune checkpoint inhibitors zalifrelimab (anti-CTLA-4) and balstilimab (anti-PD-1) in select tumors that are generally resistant to therapy.

In the Phase 1 dose escalation part of the study, the maximum tolerated dose (or maximum allowable dose) of evofosfamide in combination with zalifrelimab and balstilimab will be determined. A recommended Phase 2 dose (RP2D) will be determined based on safety and the totality of data.

The Phase 2 dose expansion part of the study will evaluate the Phase 2 dose of the triplet combination in 3 cohorts: 1) patients with locally advanced or metastatic castration-resistant prostate cancer; 2) patients with locally advanced or metastatic pancreatic cancer; and 3) patients with locally advanced or metastatic HPV-negative SCCHN. Each cohort expansion will be carried out independently.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced or metastatic castration-resistant prostate cancer, pancreatic cancer, or HPV-negative SCCHN for which no other lines of standard therapy with demonstrated clinical benefit are available or appropriate as treatment.
2. Appropriate to enter a clinical trial with a minimum estimated life expectancy of at least 3 months.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Measurable disease as defined by RECIST 1.1. Patients with castration-resistant prostate cancer can have measurable or evaluable disease per PCWG3 criteria. Patients with evaluable disease must have documented evidence of PD as defined by any of the following:

   * PSA progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least ≥4.0 ng/mL.
   * New or increasing non-bone disease per RECIST 1.1 criteria.
   * Positive bone scan with 2 or more new lesions (PCWG3).
5. Adequate bone marrow function as defined by the following laboratory test results obtained within 7 days of Cycle 1 Day 1:

   * White blood cell count ≥2500 cells/mm3.
   * Absolute neutrophil count ≥1500 cells/mm3.
   * Absolute lymphocyte count >500 cells/mm3.
   * Hemoglobin ≥9 g/dL.
   * Platelets ≥75,000 cells/mm3.
6. Adequate liver function as defined by the following laboratory test results obtained within 7 days of Cycle 1 Day 1:

   * Bilirubin ≤1.5 × institutional ULN; for patients with known Gilbert's syndrome, ≤3 × institutional ULN.
   * Aspartate aminotransferase (SGOT) and alanine aminotransferase (SGPT) ≤3 × institutional ULN; if liver metastases are present, then ≤5 × ULN is allowed.
7. At least 3 weeks from previous cytotoxic chemotherapy or radiation therapy and at least 5 half-lives or 6 weeks, whichever is shorter, from targeted or biologic therapy with the exception of CTLA-4, PD-1, or PD-L1 blocking antibodies for which only a 2 week interval is required. Patients with prostate cancer, unless they have undergone prior orchiectomy, may continue to receive androgen deprivation therapy, anti-androgen therapy, or therapy that interferes with androgenic stimulation.
8. All patients must be willing to undergo a biopsy to provide a new tumor sample within 14 days of Cycle 1 Day 1. Patients who are unable to undergo a biopsy at screening must submit archival tumor tissue retrieved within the last 6 calendar months. Patients must also consent to undergo a biopsy between Day 15 of Cycle 2 and Day 8 of Cycle 3 in those subjects which it is clinically safe and attainable. A biopsy is not required for participants with metastatic prostate cancer with bone-only disease or inaccessible soft tissue lesions.
9. Calculated creatinine clearance ≥ 60 mL/min (by the Cockcroft Gault formula) within 7 days of Cycle 1 Day 1

Exclusion Criteria:

1. A history of currently active/uncontrolled autoimmune diseases or disorders, including inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, systemic sclerosis (scleroderma), systemic lupus erythematosus, or autoimmune vasculitis (eg, Wegener's granulomatosis).
2. Patients with prior history of any Grade 3 or Grade 4 AEs from anti-CTLA-4, anti-PD-1/PD-L1, or anti-CTLA-4 and anti-PD-1/PD-L-1 combination therapy.
3. History of acute diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, abdominal carcinomatosis, or other known risk factors for bowel perforation.
4. Patients on long-term systemic steroids (>10 mg daily prednisone equivalent initiated >2 weeks prior to study enrollment). Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
5. Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study treatment hazardous or obscure the interpretation of AEs, e.g., a condition associated with frequent diarrhea or chronic skin conditions, recent surgery (within 30 days) or colonic biopsy from which the patient has not recovered, partial endocrine organ deficiencies, or substance abuse.
6. Concomitant use of QT-prolonging drugs with a risk of causing Torsades de Pointes (TdP).
7. History of risk factors for TdP, including family history of long QT syndrome.
8. Corrected QT (QTc) interval of ≥470 msec calculated according to Fridericia's formula (QTc=QT/RR [0.33]).
9. Sustained systolic blood pressure (BP) >140 mmHg or <90 mmHg and sustained diastolic BP >100 mmHg or <60 mmHg.
10. Patients with newly diagnosed, uncontrolled and/or untreated cancer-related central nervous system disease. Patients with treated brain metastases that are radiographically or clinically stable for at least 2 weeks after therapy and have no evidence of cavitation or hemorrhage in the brain lesion(s) are eligible if they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to study enrollment).
11. Uncontrolled intercurrent illness including, but not limited to, myocardial infarction within 6 months, unstable symptomatic ischemic heart disease, significant cardiac arrythmias, active uncontrolled infection requiring systemic therapy, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to study enrollment.
13. Current evidence of active and uncontrolled infection, New York Heart Association Class III-IV chronic heart failure, documented Child's class B and C cirrhosis, active symptomatic pancreatitis, or uncontrolled medical disease which, in the opinion of the investigator, could compromise assessment of study treatment efficacy.
14. Active human immunodeficiency virus infection (Exception: patients with well-controlled HIV [e.g., CD4 ≥ 350 cells/uL and undetectable viral load] who have been on an effective (drug, dosage, and schedule associated with reduction and control of the viral load) antiretroviral therapy (ART) for ≥ 4 weeks are eligible). Patients with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last 12 months are not eligible. Note: Drug-drug interactions with ART occur via many mechanisms, with cytochrome P450 CYP3A4-mediated interactions being the most common. Patients who are using concurrent strong or moderate CYP3A4 inhibitors (e.g., ritonavir, cobicistat) or strong or moderate CYP3A4 inducers must be switched to an alternate effective ART regimen ≥ 4 weeks before study enrollment or should be excluded from the study if their regimen cannot be altered.
15. Active or chronic hepatitis B or C virus infection. Patients with a history of HCV infection must have completed curative antiviral treatment and must have a viral load below the limit of quantification. A patient who is HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution is eligible.
16. Known hypersensitivity to any components of the study treatment or any of their excipients or analogs or drugs of similar chemical or biologic composition.
17. Live vaccine within 4 weeks prior to study enrollment.
18. Concomitant therapy with interleukin-2, interferon, or other non-study immunotherapy agents, or immunosuppressive agents.
19. Concomitant use of strong or moderate inhibitors or strong or moderate inducers of CYP3A4 within 14 days or 5 half-lives (whichever is longer) prior to study enrollment and for the duration of study treatment.
20. Concomitant use of anti-cancer chemotherapy, radiotherapy, hormone therapy, or targeted therapy. Patients with prostate cancer may continue treatment with anti-androgen and bone targeted therapies (e.g., zoledronic acid and denosumab). Palliative radiotherapy to nontarget lesions is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events including dose-limiting toxicities | 12 months

SECONDARY OUTCOMES:
Serious adverse events, discontinuations, and deaths | 12 months
Progression-free survival per RECIST 1.1 and iRECIST | 12 months
Objective response rate per RECIST 1.1 and iRECIST criteria (or PCWG3/RECIST for prostate cancer) | 12 months
Duration of response per RECIST 1.1 and iRECIST | 12 months
Overall survival | 12 months
Pharmacokinetic parameters including area under the concentration-time curve (AUC) for evofosfamide, Br-IPM, balstilimab, and zalifrelimab | 12 months
Pharmacokinetic parameters including Cmax for evofosfamide, Br-IPM, balstilimab, and zalifrelimab | 12 months
Pharmacokinetic parameters including t1/2 for evofosfamide, Br-IPM, balstilimab, and zalifrelimab | 12 months
Detection of anti-drug antibodies of zalifrelimab and balstilimab | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will later be determined according to ImmunoGenesis commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, ImmunoGenesis commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. Interested researchers should contact ImmunoGenesis patient-level data and supporting documents from clinical studies to conduct research.